CLINICAL TRIAL: NCT01946503
Title: Infant & Toddler Short Gut Feeding Outcomes Study
Status: Completed | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Russell Merritt, Medical Director, Nutritional Support Team and Intestinal Rehabilitation, Children's Hospital Los Angeles
Other Study IDs: CCI-13-00053
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Short Bowel Syndrome; Intestinal Failure; Home Parenteral Nutrition
Keywords: Short Gut; Short Bowel Syndrome; Intestinal Failure; Home parenteral nutrition; Feeding Behavior; Enteral Nutrition; Parent-Child Relations; Parenteral Nutrition; Digestive System Diseases
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure; Feeding Behavior; Hyperphagia; Digestive System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Short bowel syndrome: Patients followed in a clinic for short bowel syndrome
- Healthy controls: Patients seen in a general pediatric clinic without chronic or acute diseases

SUMMARY:
The purpose of this study is to better understand why children with short gut develop feeding problems.

DETAILED DESCRIPTION:
We seek to identify characteristics of our patients' histories that are associated with feeding problems in the context of availability of early prophylactic occupational therapy. We plan to review our most recent four years' experience in children with short gut syndrome with onset in early infancy who initially required home parenteral nutrition to identify risk factors or clusters of risk factors associated with food aversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in home-TPN clinic since July of 2008 with:
* Intestinal failure
* Short gut
* Onset < 3 months of age
* Received home parenteral nutrition following initial hospital discharge
* Less than 7 years of age at time of study
* Must have at least 1 parent/legal guradian willing to participate in the study

Exclusion Criteria:

* Not seen in home TPN clinic
* Short gut with onset >3 months
* No parents/legal guradians willing to participate in the study

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients seen in home-TPN clinic and subjects who meet the inclusion criteria will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Retrospective data | up to 1 year
  Data will be reviewed starting at the patient's birth. We will only be looking at patients who have been seen in the clinic since July 1, 2008; some of these will have medical records going back as early as 2006. We will continue to collect future data for up to 1 year from the beginning of data collection.

SECONDARY OUTCOMES:
Validated Questionnaires | 2 hours
  Validated questionnaires (where available) will be administered prospectively to grade current feeding competence for age, assess developmental status, assess food preferences and score parental stress. Only the food preference questionnaire will be administered to the healthy control group.

CONTACTS AND LOCATIONS:
Overall Officials: Russell J Merritt, MD, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bazyk S. Factors associated with the transition to oral feeding in infants fed by nasogastric tubes. Am J Occup Ther. 1990 Dec;44(12):1070-8. doi: 10.5014/ajot.44.12.1070. PMID 2126165
- [Background] Black MM, Aboud FE. Responsive feeding is embedded in a theoretical framework of responsive parenting. J Nutr. 2011 Mar;141(3):490-4. doi: 10.3945/jn.110.129973. Epub 2011 Jan 26. PMID 21270366
- [Background] Byars KC, Burklow KA, Ferguson K, O'Flaherty T, Santoro K, Kaul A. A multicomponent behavioral program for oral aversion in children dependent on gastrostomy feedings. J Pediatr Gastroenterol Nutr. 2003 Oct;37(4):473-80. doi: 10.1097/00005176-200310000-00014. PMID 14508219
- [Background] Davies WH, Satter E, Berlin KS, Sato AF, Silverman AH, Fischer EA, Arvedson JC, Rudolph CD. Reconceptualizing feeding and feeding disorders in interpersonal context: the case for a relational disorder. J Fam Psychol. 2006 Sep;20(3):409-17. doi: 10.1037/0893-3200.20.3.409. PMID 16937997
- [Background] Engstrom I, Bjornestam B, Finkel Y. Psychological distress associated with home parenteral nutrition in Swedish children, adolescents, and their parents: preliminary results. J Pediatr Gastroenterol Nutr. 2003 Sep;37(3):246-50. doi: 10.1097/00005176-200309000-00008. PMID 12960644
- [Background] Geertsma MA, Hyams JS, Pelletier JM, Reiter S. Feeding resistance after parenteral hyperalimentation. Am J Dis Child. 1985 Mar;139(3):255-6. doi: 10.1001/archpedi.1985.02140050049020. PMID 3919567
- [Background] Lacaille F, Vass N, Sauvat F, Canioni D, Colomb V, Talbotec C, De Serre NP, Salomon J, Hugot JP, Cezard JP, Revillon Y, Ruemmele FM, Goulet O. Long-term outcome, growth and digestive function in children 2 to 18 years after intestinal transplantation. Gut. 2008 Apr;57(4):455-61. doi: 10.1136/gut.2007.133389. Epub 2007 Dec 13. PMID 18079282
- [Background] Gottrand F, Staszewski P, Colomb V, Loras-Duclaux I, Guimber D, Marinier E, Breton A, Magnificat S. Satisfaction in different life domains in children receiving home parenteral nutrition and their families. J Pediatr. 2005 Jun;146(6):793-7. doi: 10.1016/j.jpeds.2005.01.034. PMID 15973321
- [Background] Pedersen SD, Parsons HG, Dewey D. Stress levels experienced by the parents of enterally fed children. Child Care Health Dev. 2004 Sep;30(5):507-13. doi: 10.1111/j.1365-2214.2004.00437.x. PMID 15320927
- [Background] Wilken M. The impact of child tube feeding on maternal emotional state and identity: a qualitative meta-analysis. J Pediatr Nurs. 2012 Jun;27(3):248-55. doi: 10.1016/j.pedn.2011.01.032. Epub 2011 Mar 15. PMID 22525813